CLINICAL TRIAL: NCT05870488
Title: iFuse TORQ for the Treatment of Sacroiliac Joint Dysfunction
Acronym: STACI
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: SI-BONE, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 301140
Record Dates: First submitted 2023-05-12; First posted 2023-05-23 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Sacroiliac Joint Dysfunction; Sacroiliac; Fusion; Sacroiliac Disorder; Sacroiliac Joint Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Use of iFuse TORQ for SI Joint Fusion (Other): Participants with SI joint dysfunction are treated with iFuse TORQ.
  Interventions: Device: Use of iFuse TORQ

INTERVENTIONS:
Device: Use of iFuse TORQ — Use of iFuse TORQ for the treatment of SI Joint dysfunction

SUMMARY:
iFuse TORQ for the Treatment of Sacroiliac Joint Dysfunction (STACI) is a prospective, multicenter, study of SIJ fusion using the iFuse TORQ implant system.

DETAILED DESCRIPTION:
This trial is a prospective, multicenter, study of SIJ fusion using the iFuse TORQ implant system. The goal of the trial is to demonstrate the effectiveness of the device for its intended use.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 21 at time of screening
2. Patient has lower back / buttock pain for at least 6 months inadequately responsive to non-surgical care
3. Diagnosis of sacroiliac joint dysfunction (degenerative sacroiliitis or sacroiliac disruption)
4. Baseline Oswestry Disability Index (ODI) score of at least 30%
5. Baseline SIJ pain score of at least 5 on 0-10 numerical rating scale
6. BMI < 35
7. Patient has signed study-specific informed consent form

Exclusion Criteria:

1. ASA score 4 or 5
2. Severe back pain due to other causes, such as lumbar disc degeneration, lumbar disc herniation, lumbar spondylolisthesis, lumbar spinal stenosis, lumbar facet degeneration, and lumbar vertebral body fracture
3. Other known sacroiliac pathology such as: inflammatory sacroiliitis (e.g., ankylosing spondylitis or other HLA-associated spondyloarthropathy), tumor, infection, acute fracture
4. Cluneal neuralgia
5. Previous SIJ implant placement, including allograft
6. Anatomic anomalies/defects that would preclude safe and/or biomechanically acceptable device placement
7. History of recent (<1 year) major trauma to pelvis
8. Previously diagnosed or suspected severe osteoporosis (defined as prior T-score < -2.5 or history of osteoporotic fracture).
9. Chronic rheumatologic condition (e.g., rheumatoid arthritis)
10. Current diagnosis of fibromyalgia
11. Known allergy to titanium or titanium alloys
12. Current local or systemic infection that raises the risk of surgery
13. Patient currently receiving or seeking worker's compensation, disability remuneration, and/or involved in injury litigation
14. Currently pregnant or planning pregnancy in the next 2 years (self-reported)
15. Patient is a prisoner or a ward of the state.
16. Known or suspected active drug or alcohol abuse, including opioids
17. Diagnosed psychiatric disease (e.g., schizophrenia, major depression, personality disorders) that could interfere with study participation
18. Currently participating in another interventional clinical trial

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2025-04-23 (Actual); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Change in SI joint pain measured by numerical rating scale (NRS) | At baseline and 6 months
  Change in SI joint pain measured by NRS (0- no pain to 10- worst pain imaginable)

SECONDARY OUTCOMES:
Improvement from baseline in SI joint (SIJ) pain | At baseline, 1-, 3-, 6-, 12-, and 24-months
  Improvement from baseline in SIJ pain as measured by numeric rating scale (0- no pain to 10- worst pain imaginable).
Improvement from baseline in disability | At baseline, 1-, 3-, 6-, 12-, and 24-months
  Improvement from baseline in disability as measured by Oswestry Disability Index
Improvement from baseline in quality of life | At baseline, 1-, 3-, 6-, 12-, and 24-months
  Improvement from baseline in aggregate quality of life and individual domains as measured by PROMIS-29.
Proportion of subjects with a complication rated as probably or definitely related to the procedure or device. | At baseline, 1-, 3-, 6-, 12-, and 24-months
Evidence of bone binding | At baseline and 24 months
  Evidence of bone binding to at least 50% of the porous surface area of each implanted device
Proportion of treated sides showing signs of loosening of iFuse TORQ or other instrumentation | At baseline and 24 months
  Proportion of treated sides showing signs of loosening of iFuse TORQ or other instrumentation, as evidenced by both radiopaque areas around implant plus bony reaction ("rind") near implant
Proportion of iFuse TORQ implants that show evidence of device migration | At baseline and 24 months
Proportion of iFuse TORQ implants that show breakage | At baseline and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Stacie Tran, MPH, Study Director — SI-BONE
Locations (14):
- United States (14):
  - Napa Valley Orthopaedics, Napa, California
  - Source Healthcare, Santa Monica, California
  - Comprehensive Pain and Spine Specialists, Shelbyville, Indiana
  - Ascentist Healthcare, Leawood, Kansas
  - Crimson Pain Management, Overland Park, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Clearway Pain, Annapolis, Maryland
  - St Louis Pain Consultants, Chesterfield, Missouri
  - Nevada Advanced Pain, Reno, Nevada
  - Clinical Investigations, Edmond, Oklahoma
  - Neurological Associates of Lancaster, Lancaster, Pennsylvania
  - Advanced Pain Institute of Texas, Lewisville, Texas
  - Anesis Spine & Pain Care, Renton, Washington
  - Pro Spine and Pain, Milwaukee, Wisconsin